CLINICAL TRIAL: NCT06293560
Title: Microphthalmia, Anophthalmia, and Coloboma Genetic Epidemiology in Children
Acronym: MAGIC
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Eye Institute (NEI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Philip J Lupo, Principal Investigator, Professor of Pediatrics; Director, Epidemiology and Population Sciences Program, Baylor College of Medicine
Other Study IDs: H-49046; 5U01EY032403-03 (NIH)
Record Dates: First submitted 2024-02-21; First posted 2024-03-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Microphthalmia; Coloboma; Anophthalmia
MeSH Terms: conditions — Microphthalmos; Coloboma; Anophthalmos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The investigators are inviting families to take part in a research study that will help us better understand the physical characteristics associated with children who have Microphthalmia, Anophthalmia, and Coloboma (MAC) and how changes in their DNA sequence, called genetic mutations, play a role in the risk of developing MAC

DETAILED DESCRIPTION:
This study is focused on gathering data on individuals diagnosed with some of the more common visually threatening congenital eye defects collectively referred to as MAC complex; anophthalmia (total absence of the globe), microphthalmia (anomalously small eye in the orbit), and coloboma (failure of the closure of the fetal fissure).

Our long-term goal is to improve prevention efforts for and clinical management of MAC. The objectives of the current study are to 1) better define the MAC phenotype and 2) characterize the role of known and newly identified pathogenic genetic variants that confer MAC susceptibility.

To do this, the investigators are leveraging resources to identify MAC cases through the Texas Birth Defects Registry (TBDR), Texas Children's Hospital (TCH), and through direct referrals from our study partners. The investigators intend to conduct secondary analyses by leveraging the existing collaborative relationship with the New York State Newborn Screening Program (NYSNSP). Also, the investigators are utilizing the resources of the National Institutes of Health (NIH) Clinical Center to comprehensively phenotype cases with MAC, and the National Eye Institute (NEI) Ophthalmic Genomics Laboratory to identify genetic variants underlying MAC phenotypes.

ELIGIBILITY:
Inclusion Criteria:

1. All MAC cases
2. Parents of the above children.
3. Siblings of the above children.
4. English or Spanish speaking.

Exclusion Criteria:

All subjects who do not meet the inclusion criteria listed above.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children diagnosed with congenital microphthalmia, anophthalmia, or coloboma (without a recognized syndrome).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-09-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Stage 1 | End of study, on or before 12/31/2032
  We are conducting interviews to collect detailed pregnancy, medical and family histories; review medical records to identify cases with chromosomal abnormalities or other syndromic diagnosis (that were not identified by the TBDR) and associated malformations, as well as to assess clinical course; and collect saliva samples that may be used to extract DNA to be analyzed for genetic mutations.
Stage 2 | End of study, on or before 12/31/2032
  We are also conducting in-person, virtual, or remote physical assessments to obtain detailed phenotypic information including three-dimensional (3D) digital imaging to capture facial phenotype of cases and their parents. We also collect blood samples during this stage.
Stage 3 | End of study, on or before 12/31/2032
  We are working closely with collaborators at the NIH Clinical Center to conduct deep phenotyping of children with MAC, who do not have a diagnosed syndrome, as well as their first-degree family members. This may include complete eye examinations, neuropsychological testing, hearing evaluation, additional facial imaging, echocardiograms, and magnetic resonance imaging (MRI) of the brain.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Langlois PH, Marengo L, Lupo PJ, Drummond-Borg M, Agopian AJ, Nembhard WN, Canfield MA. Evaluating the proportion of isolated cases among a spectrum of birth defects in a population-based registry. Birth Defects Res. 2023 Jan 1;115(1):21-25. doi: 10.1002/bdr2.1990. Epub 2022 Feb 26. PMID 35218607
- [Background] Selzer EB, Blain D, Hufnagel RB, Lupo PJ, Mitchell LE, Brooks BP. Review of evidence for environmental causes of uveal coloboma. Surv Ophthalmol. 2022 Jul-Aug;67(4):1031-1047. doi: 10.1016/j.survophthal.2021.12.008. Epub 2021 Dec 31. PMID 34979194
- [Background] Schraw JM, Benjamin RH, Scott DA, Brooks BP, Hufnagel RB, McLean SD, Northrup H, Langlois PH, Canfield MA, Scheuerle AE, Schaaf CP, Ray JW, Chen H, Swartz MD, Mitchell LE, Agopian AJ, Lupo PJ. A Comprehensive Assessment of Co-occurring Birth Defects among Infants with Non-Syndromic Anophthalmia or Microphthalmia. Ophthalmic Epidemiol. 2021 Oct;28(5):428-435. doi: 10.1080/09286586.2020.1862244. Epub 2020 Dec 20. PMID 33345678